CLINICAL TRIAL: NCT01649388
Title: A Single-arm, Multi-center, Exploratory Safety and Efficacy Study of FCR001 Cell-based Therapy to Induce Donor-specific Tolerance in Previously Transplanted Recipients of a Kidney From a Living Donor, and Safety in FCR001 Donors
Brief Title: A Safety and Efficacy Study of FCR001 Cell Therapy in Previously Transplanted Living Donor Kidney Recipients
Acronym: FREEDOM-2
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: study terminated by sponsor
Sponsor: Talaris Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FCR001B2201
Record Dates: First submitted 2012-06-29; First posted 2012-07-25 (Estimated); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Kidney Transplantation
Keywords: Selective allograft tolerance; Stem cell therapy; Living donor kidney transplant; Immune tolerance; Durable chimerism; Immunosuppression; Immunosuppressive medications; Organ transplant rejection; Anti-rejection medications

STUDY DESIGN:
Intervention Model Description: approximately 15 Donor/Recipient pairs
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- FCR001 (Experimental): Recipients 3-12 months post-living kidney transplantation undergo non-myeloablative conditioning followed by infusion of an enriched hematopoietic stem cell product derived from the same living donor's peripheral blood stem cells
  Interventions: Biological: FCR001

INTERVENTIONS:
Biological: FCR001 — Enriched hematopoietic stem cell infusion

SUMMARY:
An open-label study to assess the safety, tolerability, and efficacy of FCR001 cell therapy in adult recipients 3-12 months after kidney transplantation from a living donor.

DETAILED DESCRIPTION:
The purpose of this study is to assess the safety, tolerability, preliminary efficacy, and overall benefit of FCR001 cell therapy in previously transplanted recipients of a kidney from a living donor.

FCR001 is a novel, cryopreserved allogeneic somatic cell therapy, derived from mobilized peripheral blood mononuclear cells from the same donor as the allograft, and containing hematopoietic progenitor cells, facilitating cells, and αβ T cells. The rationale is to establish durable chimerism and donor-specific tolerance in the recipient enabling freedom from chronic immunosuppression (IS) and its associated toxicities.

ELIGIBILITY:
Main Inclusion Criteria:

1. Recipient age ≥18 years old.
2. Donor age ≥18 and ≤60 years old at the time of signing informed consent.
3. Recipient of a first kidney transplant from a living donor 3-12 months prior to signing informed consent.
4. Stable renal allograft function ≥60 mL/min/1.73m^2 prior to screening (defined as <25% decrease in eGFR (by Modification of Diet in Renal Disease formula [MDRD4]) between the last 2 consecutive visits and per investigator judgment).
5. Donor between 3 weeks and 12 months after kidney donation, willing to undergo mobilization, apheresis, and 12-month safety follow-up.

Main Exclusion Criteria (Recipient and Donor):

1. Donor/recipient crossmatch positive at time of living donor kidney transplantation.
2. Recipient or donor with use of other investigational drugs within 30 days (or within 5 drug half-lives) of signing informed consent.
3. Recipient or donor with history of hypersensitivity to any of the study drugs or drugs of similar chemical classes.
4. Recipient and donor who are identical twins.
5. Pregnant or nursing (lactating) woman.
6. Recipient or donor with history of malignancy or premalignant syndrome (e.g., myelodysplastic syndrome, monoclonal gammopathy of renal significance [MGRS], monoclonal gammopathy of unknown significant [MGUS]) of any organ system (other than localized excised non-melanomatous lesions of the skin or in-situ cervical cancer), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
7. Recipient or donor with known bone marrow aplasia.

   Main Exclusion Criteria (Recipient-Only):
8. Multi-organ or cell transplant recipient.
9. Blood type ABO incompatible with donor.
10. Positive donor-specific antibody (DSA) at any time pre- or post-transplant (to be confirmed within 30 days prior to FCR001 infusion).
11. Panel Reactive Antibodies (PRA) >80% at the time of living donor kidney transplantation.
12. Induction with alemtuzumab at the time of living donor kidney transplantation.
13. History of acute rejection (biopsy-proven or suspected and treated) or recurrent kidney disease following living donor kidney transplantation.
14. Findings consistent with acute rejection or recurrent disease on the Screening biopsy.
15. Demonstrated intolerance to maintenance immunosuppression with tacrolimus and MMF or MPS.
16. Being maintained on oral corticosteroids (prednisone >10 mg/day or equivalent).
17. Positive for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV). Recipients with history of HCV infection may participate if there is a documented history of treatment with an anti-HCV agent and either one (1) documented negative PCR at least three (3) months after last dose of treatment, or two (2) documented negative PCRs at least 2 weeks apart over a maximum of 4 weeks.
18. Positive for BKV, CMV, or EBV by PCR at screening.
19. Having any baseline condition requiring or anticipated to require chronic or intermittent use of systemic steroids or other IS (e.g., autoimmune disease, asthma) throughout the course of the study.
20. Having a body mass index (BMI) < 18 or > 35 kg/m^2.
21. Requiring systemic anticoagulation, (e.g., for hypercoagulation disorders, deep vein thrombosis, atrial fibrillation) that cannot be temporarily interrupted with would preclude renal biopsy.
22. Having contraindication to TBI according to local radiologist.
23. History of autologous or allogeneic hematopoietic progenitor or mesenchymal stem cell transplant prior to signing informed consent.

    Main Exclusion Criteria (Donor-Only):
24. Biologically unrelated (i.e., no genetic relationship) female donor transplant to male recipient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-10-15 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Proportion of FCR recipients (FCR-R) who are free from immunosuppression (IS), without biopsy-proven acute rejection (BPAR), at 24 months post-FCR001 infusion | From infusion to 24 months

SECONDARY OUTCOMES:
Change in renal function (estimated Glomerular Filtration Rate [eGFR] by Modification of Diet in Renal Disease [MDRD4]) from baseline (Day 1, prior to FCR001 infusion) to Month 24 in FCR recipients | From Day 1 prior to infusion to 24 months
Renal allograft function (eGFR by MDRD4) | From infusion to 24 months and 60 months
Change in renal allograft function over time by MDRD4 | From infusion to 24 months and 60 months
Renal allograft function (eGFR) by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula | From infusion to 24 months and 60 months
Change in renal allograft function over time by CKD-EPI | From infusion to 24 months and 60 months
Time to event for the composite of BPAR, renal graft loss, death, or lost to follow-up and each component | From infusion to 60 months
Incidence of composite endpoint of BPAR, renal graft loss, or death | From infusion to 12 months, 24 months and 60 months
Incidence and severity of adverse events (AEs), serious adverse events (SAEs), and AEs leading to study and/or regimen discontinuation | From informed consent to 12 months, 24 months and 60 months
Incidence of BK viremia, viruria, infection, and nephropathy | From informed consent to 12 months, 24 months and 60 months
Incidence of donor chimerism by visit | From infusion to 60 months
Incidence of acute and chronic GvHD | From infusion to 60 months
Incidence of engraftment syndrome | From infusion to 60 months
Incidence of recipient autologous apheresis product infusion | From infusion to 60 months
Renal graft survival for recipients transiently chimeric | From infusion to 60 months
Incidence of composite endpoint of BPAR, death, renal graft loss, or lost to follow-up in FCR-R who did not achieve durable chimerism or able to wean or remain off IS | From infusion to 60 months

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Minnesota Medical Center, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No